CLINICAL TRIAL: NCT02931188
Title: A Cross-sectional REVEAL Sub-study Evaluating the Effect of Anacetrapib on Vascular Function and Arterial Stiffness [An Investigator Led Sub-study of HPS3/TIMI 55: REVEAL]
Brief Title: The Effect of Anacetrapib on Vascular Function and Arterial Stiffness
Acronym: REVEAL-Vasc
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: British Heart Foundation Cambridge Centre of Excellence (Unknown)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Clinical Pharmacologist & Physician/Associate Lecturer, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: REVEAL-Vasc
Record Dates: First submitted 2016-09-12; First posted 2016-10-12 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Atherosclerotic Cardiovascular Disease; Vascular Disease
Keywords: Vascular Diseases; Lipids; Cholesteryl Ester Transfer Protein (CETP) Inhibition; Anacetrapib; Cardiovascular Disease; Cholesterol
MeSH Terms: conditions — Atherosclerosis; Vascular Diseases; Inhibition, Psychological; Cardiovascular Diseases | interventions — anacetrapib; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 15ml blood samples will be collected from each participant at visit 1.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anacetrapib: Participants who received anacetrapib, in addition to statin on the HPS3/TIMI 55: REVEAL trial.
  Interventions: Drug: Anacetrapib; Drug: Statin
- Placebo: Participants who received placebo, in addition to statin on the HPS3/TIMI 55: REVEAL trial.
  Interventions: Drug: Statin; Drug: Placebo

INTERVENTIONS:
Drug: Anacetrapib — No drug administration will occur on this sub-study. Participants will receive treatment on the main trial HPS3/TIMI 55: REVEAL (NCT01252953)
  Groups: Anacetrapib
Drug: Statin — No drug administration will occur on this sub-study. Participants will receive treatment on the main trial HPS3/TIMI 55: REVEAL (NCT01252953)
Drug: Placebo — No drug administration will occur on this sub-study. Participants will receive treatment on the main trial HPS3/TIMI 55: REVEAL (NCT01252953)
  Groups: Placebo

SUMMARY:
There are currently no studies evaluating the effect of anacetrapib on blood vessel function and stiffness of the arteries. The REVEAL-Vasc trial will assess whether anacetrapib, in addition to atorvastatin (LDL-C lowering drug) treatment, results in greater endothelial-dependent vascular function and aortic stiffness in patients with established cardiovascular disease, compared to adding placebo.

Participants will be asked to provide a blood sample and pulse Wave Velocity/Pulse Wave Analysis and Flow Mediated Dilation will be carried out to assess blood vessel function and stiffness of the arteries. REVEAL-Vasc is an investigator led sub-study of HPS3/TIMI 55: REVEAL (Randomized Evaluation of the Effects of Anacetrapib through Lipid modification): A large-scale, randomized placebo-controlled trial of the clinical effects of anacetrapib among people with established vascular disease (NCT01252953) which is coordinated by OXFORD CTSU.

No treatment will be received on this sub-study, therefore only participants who have been enrolled in HPS3/TIMI55 REVEAL in which participants received anacetrapib with atorvastatin or placebo will be considered for this trial.

DETAILED DESCRIPTION:
REVEAL-Vasc is an investigator led sub-study of HPS3/TIMI 55: REVEAL. Participants who previously enrolled on HPS3/TIMI 55: REVEAL and received treatment will be invited to participate in this sub-study. Participants will attend a screening and an assessment visit during which Pulse Wave Velocity/ Pulse Wave Analysis and Flow Mediated Dilation will be carried out to assess blood vessel function and stiffness. A blood sample will also be taken from participant to assess CRP and lipid profile. Since participants will have received treatment on the main trial HPS3/TIMI 55: REVEAL, no treatment will be received on this sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been randomised into the HPS3/TIMI 55- REVEAL study (NCT01252953)

Exclusion Criteria:

* Any concomitant condition that, at the discretion of the investigator, may affect the participant's ability to complete the study or study procedures
* Atrial fibrillation at time of assessment
* Inability to provide informed consent
* Inability to refrain from caffeine containing products for 6 hours prior to study visit
* Inability to refrain from smoking for 2 hours prior to study visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this sub-study will be recrited from the HPS3/TIMI 55- REVEAL trial (NCT01252953).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The effect of treatment on flow-mediated dilation (FMD) | Visits 0-1 (day 0 up to approximately day 28 depending on scheduling of visits)
  Measured by FMD as a surrogate measure of endothelial-dependent vasodilation

SECONDARY OUTCOMES:
The effect of treatment on aortic (carotid-to-femoral) Pulse Wave Velocity (PWV) | Visits 0-1 (day 0 up to approximately day 28 depending on scheduling of visits)
  Measured by PWV as a surrogate measure of aortic stiffness
The effect of treatment on central blood pressure | Visits 0-1 (day 0 up to approximately day 28 depending on scheduling of visits)
  As a measure of central haemodynamics
The effect of treatment on sublingual glyceryl trinitrate (GTN) response on artery dilation | Visits 0-1 (day 0 up to approximately day 28 depending on scheduling of visits)
  Measured by FMD as a surrogate measure of endothelial-independent vasodilation

OTHER OUTCOMES:
The analysis of low density lipoproteins, high density lipoproteins, total cholesterol and triglycerides (amongst other analytes) from collected blood samples | Visits 0-1 (day 0 up to approximately day 28 depending on scheduling of visits)
  As a measure of treatment on lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB, MA, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Clinical Investigation Ward, Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: REVEAL main trial clinicaltrials.gov record — https://clinicaltrials.gov/ct2/show/NCT01252953?term=NCT01252953&rank=1